CLINICAL TRIAL: NCT01061411
Title: Phase I Study of Dalteparin, A Low Molecular Weight Heparin (LMWH), in Combination With Sunitinib (SU11248), an Oral, Selective Multi-targeted Tyrosine Kinase Inhibitor, as First Line Treatment, in Patients With Metastatic Renal Cell Carcinoma
Brief Title: Dalteparin and Sunitinib Malate as First-Line Therapy in Treating Patients With Kidney Cancer That is Metastatic or Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 145508; NCI-2009-01694 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 145508 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2010-02-01; First posted 2010-02-03 (Estimated); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Clear Cell Sarcoma of the Kidney; Recurrent Renal Cell Carcinoma; Stage III Renal Cell Cancer; Stage IV Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Dalteparin; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (sunitinib malate, dalteparin) (Experimental): Patients receive sunitinib malate PO QD in weeks 1-4 and dalteparin SC QD in week 6 during course 1. In all subsequent courses, patients receive sunitinib malate PO QD in weeks 1-4 and dalteparin SC QD in weeks 1-6. Courses repeat every 6 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Dalteparin; Other: Pharmacological Study; Drug: Sunitinib Malate

INTERVENTIONS:
Drug: Dalteparin — Given SC
Other: Pharmacological Study — Correlative studies
Drug: Sunitinib Malate — Given PO
  Other Names: SU011248; SU11248; sunitinib; Sutent

SUMMARY:
This phase I trial studies the side effects and best dose of dalteparin when given together with sunitinib malate in treating patients with kidney cancer that has spread to other parts of the body or cannot be removed by surgery. Anticoagulants, such as dalteparin, help prevent blood clots and have been shown to increase survival in patients with cancer. Anticoagulants may also prevent the formation of new blood vessels. Sunitinib malate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by inhibiting new blood vessels and blocking blood flow to the tumor. Giving dalteparin together with sunitinib malate may starve tumors and kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the recommended dosing for the combination of sunitinib (sunitinib malate) and dalteparin in patients with metastatic renal cell carcinoma.

II. To evaluate safety and tolerability for the combination of sunitinib and dalteparin in patients with metastatic renal cell carcinoma.

III. To determine early signs of clinical activity of the combination of sunitinib and dalteparin in patients with metastatic renal cell carcinoma.

SECONDARY OBJECTIVES:

I. To determine the clinical response rate of sunitinib and dalteparin in patients with metastatic renal cell carcinoma.

II. To determine time-to-progression (TTP) and overall survival amongst patients with metastatic renal cell carcinoma receiving sunitinib and dalteparin.

III. To determine the effect of sunitinib alone and dalteparin alone compared to the combination of dalteparin plus sunitinib on plasma coagulation parameters.

IV. To determine the effect of sunitinib alone and dalteparin alone compared to the combination of dalteparin plus sunitinib on angiogenesis parameters in blood.

OUTLINE: This is a dose-escalation study of dalteparin.

Patients receive sunitinib malate orally (PO) once daily (QD) in weeks 1-4 and dalteparin subcutaneously (SC) QD in week 6 during course 1. In all subsequent courses, patients receive sunitinib malate PO QD in weeks 1-4 and dalteparin SC QD in weeks 1-6. Courses repeat every 6 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 4 weeks and then every 3 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed renal cell carcinoma that is metastatic or unresectable
* Renal carcinoma patients with predominant clear-cell histology are eligible; papillary renal cell carcinoma, oncocytoma, collecting duct tumors and transitional cell carcinoma are NOT eligible
* No prior systemic treatments for metastatic disease are permitted, including antiangiogenic therapy, immunotherapy, chemotherapy and investigational therapy
* Prior palliative radiation to metastatic lesion(s) is permitted, provided there is at least one measurable and/or evaluable lesion(s) that has not been irradiated
* Radiation therapy must be completed > 4 weeks prior to registration
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension as >= 20 mm with conventional techniques or as approximately >= 10 mm with spiral computed tomography (CT) scan (Response Evaluation Criteria in Solid Tumors [RECIST] 1.0 criteria)
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Leukocytes > 3,000/mm^3
* Absolute neutrophil count > 1,500/mm^3
* Platelets > 100,000/mm^3
* Total bilirubin < 1.5 x laboratory upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/ alanine transaminase (ALT) (serum glutamate pyruvate transaminase [SGPT]) < 2.5 x laboratory ULN
* Creatinine < 1.5 x laboratory ULN
* Prothrombin time (PT)/international normalized ratio (INR) < 1.5
* Urine protein < 1+; if > 1+, 24 hour urine protein should be obtained and should be < 1000 mg
* Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation
* Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document
* Except for Dalteparin that will be administered as a study drug, the patients should not take any other anticoagulants or antiplatelet agents during the study, including but not limited to nonsteroidal anti-inflammatory drugs (NSAID) (any dose of aspirin), warfarin or other anticoagulants

Exclusion Criteria:

* Patients may not be receiving any other investigational agents
* Patients with known central nervous system (CNS) metastases; patients should have a head CT/magnetic resonance imaging (MRI) within 4 weeks prior to treatment initiation; any imaging abnormality indicative of CNS metastases will exclude the patient from the study
* Patients with a "currently active" second malignancy other than non-melanoma skin cancers are not eligible; patients are not considered to have a "currently active" malignancy if they have completed anti-cancer therapy and are considered by their physician to be at less than 30% risk of relapse
* Patients with a large (> 2 cm) pulmonary lesion involving the trachea or one of the main bronchus and any endobronchial lesion
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to dalteparin
* Evidence of bleeding diathesis within last 6 months
* Serious or non-healing wound, ulcer or bone fracture or active peptic ulceration
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure (New York Association class II, III, or IV), angina pectoris requiring nitrate therapy, recent myocardial infarction (< the last 6 months), cardiac arrhythmia, history of cerebrovascular accident (CVA) within 6 months (thrombotic or hemorrhagic), hypertension (defined as blood pressure of > 160 mmHg systolic and/or > 90 mm Hg diastolic on medication), hemorrhagic retinopathy, history of peripheral vascular disease, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients with an ejection fraction < 50% by multi gated acquisition scan (MUGA) scan are not eligible
* Pregnant women are excluded from this study
* History of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 28 days prior to day 1 therapy
* Invasive procedures defined as:

  * Major surgical procedure, open biopsy, or significant traumatic injury within 6 weeks prior to day 1 therapy
  * Anticipation of need for major surgical procedures during the course of the study
  * Core biopsy within 7 days prior to start therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-02-06 (Actual); Primary Completion 2015-10-14 (Actual); Study Completion 2017-04-21 (Actual)

PRIMARY OUTCOMES:
Early signs of clinical activity of the combination of sunitinib malate and dalteparin | Up to 4 years
Incidence of toxicities for the combination of dalteparin and sunitinib malate | Up to 4 weeks after last treatment
  Toxicities will be summarized by tabulation. Summaries will be made across all types of toxicities and by grade and type.
Recommended dosing for the combination of dalteparin and sunitinib malate | Up to 4 weeks
  The maximally tolerated dose (MTD) will be the highest dose at which < 33% of patients (=< 2 out of 6 patients) suffer from dose limiting toxicities (DLTs) related to the combination treatment.

SECONDARY OUTCOMES:
Clinical response rate of dalteparin and sunitinib malate, determined as the proportion of treated patients who had partial or complete response according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.0 | Up to 4 weeks after last treatment
Overall survival | Up to 4 years
  Described in all patients using Kaplan-Meier curves.
TTP | Up to 4 years
  Described in all patients using Kaplan-Meier curves.

OTHER OUTCOMES:
Changes in angiogenesis parameters in blood | Baseline to 4 weeks after last treatment
  Each will be explored to determine if transformations (e.g. log or square-root) are necessary to achieve normality. For each of baseline and changes, exploratory plots (e.g. histograms, boxplots) will be created and means will be estimated along with 95% confidence intervals. Wilcoxon signed-rank tests will be used to determine whether or not the data shows evidence of changes from baseline.
Changes in plasma coagulation parameters | Baseline to 4 weeks after last treatment
  Each will be explored to determine if transformations (e.g. log or square-root) are necessary to achieve normality. For each of baseline and changes, exploratory plots (e.g. histograms, boxplots) will be created and means will be estimated along with 95% confidence intervals. Wilcoxon signed-rank tests will be used to determine whether or not the data shows evidence of changes from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Saby George, Principal Investigator — Roswell Park Cancer Institute
Locations (4):
- United States (2):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Roswell Park Cancer Institute, Buffalo, New York
- Netherlands (2):
  - Academ Zienkenhuis Bij De University, Amsterdam
  - VU University Medical Center, Amsterdam